CLINICAL TRIAL: NCT03748979
Title: A 3-Part, Randomized, Double-Blind, Placebo-Controlled, Multiple Rising Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TAK-925 in Healthy Volunteers and Patients With Narcolepsy
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TAK-925 in Healthy Volunteers and Participants With Narcolepsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-925-1003; U1111-1221-3144 (Other: WHO); JapicCTI-184207 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-11-15; First posted 2018-11-21 (Actual); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Healthy Participants; Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — TAK-925

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (17):
- Cohort A1; TAK-925 (Dose Level A1) (Experimental): TAK-925, Dose Level A, once daily for up to 7 days in healthy participants.
  Interventions: Drug: TAK-925
- Cohort A2; TAK-925 (Dose Level A2) (Experimental): TAK-925, Dose Level A2, once daily for up to 7 days in healthy participants. Dose level will be determined based on the data of safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TAK-925
- Cohort A3; TAK-925 (Dose Level A3) (Experimental): TAK-925, Dose Level A3, once daily for up to 7 days in healthy participants. This group is an additional optional cohort and dose level will be determined based on the data of safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TAK-925
- Cohort A4; TAK-925 (Dose Level A4) (Experimental): TAK-925, Dose Level A4, once daily for up to 7 days in healthy participants. This group is an additional optional cohort and dose level will be determined based on the data of safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TAK-925
- Cohort A5; TAK-925 (Dose Level A5) (Experimental): TAK-925, Dose Level A5, once daily for up to 7 days in healthy participants. This group is an additional optional cohort and dose level will be determined based on the data of safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TAK-925
- Cohort A6; TAK-925 (Dose Level A6) (Experimental): TAK-925, Dose Level A6, once daily for up to 7 days in healthy elderly participants. This group is an additional optional cohort and dose level will be determined based on the data of safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TAK-925
- Part A (Cohorts A1-A6); TAK-925 Placebo (Placebo Comparator): TAK-925 Placebo, once daily for up to 7 days in healthy participants.
  Interventions: Drug: Placebo
- Cohort B1; TAK-925 (Dose Level B1) (Experimental): TAK-925, Dose Level B1, once daily for up to 7 days in participants with narcolepsy.
  Interventions: Drug: TAK-925
- Cohort B2; TAK-925 (Dose Level B2) (Experimental): TAK-925, Dose Level B2, once daily for up to 7 days in participants with narcolepsy. Dose level will be determined based on the data of safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TAK-925
- Cohort B3; TAK-925 (Dose Level B3) (Experimental): TAK-925, Dose Level B3, once daily for up to 7 days in participants with narcolepsy. This group is an additional optional cohort and dose level will be determined based on the data of safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TAK-925
- Cohort B4; TAK-925 (Dose Level B4) (Experimental): TAK-925, Dose Level B4, once daily for up to 7 days in participants with narcolepsy. This group is an additional optional cohort and dose level will be determined based on the data of safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TAK-925
- Part B (Cohorts B1-B4); TAK-925 Placebo (Placebo Comparator): TAK-925 Placebo, once daily for up to 7 days in participants with narcolepsy.
  Interventions: Drug: Placebo
- Cohort C1; TAK-925 (Dose Level C1) (Experimental): TAK-925, Dose Level C1, once daily for up to 7 days in participants with narcolepsy. Dose level will be determined based on the data of safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TAK-925
- Cohort C2; TAK-925 (Dose Level C2) (Experimental): TAK-925, Dose Level C2, once daily for up to 7 days in participants with narcolepsy. This group is an additional optional cohort and dose level will be determined based on the data of safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TAK-925
- Part C (Cohorts C1-C2); TAK-925 Placebo (Placebo Comparator): TAK-925 Placebo, once daily for up to 7 days in participants with narcolepsy.
  Interventions: Drug: Placebo
- Cohort A'1; TAK-925 (Dose Level A'1) (Experimental): TAK-925, Dose Level A'1, single dose in healthy participants.
  Interventions: Drug: TAK-925
- Cohort A'2; TAK-925 (Dose Level A'2) (Experimental): TAK-925, Dose Level A'2, single dose in healthy participants. Dose level will be determined based on the data of safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TAK-925

INTERVENTIONS:
Drug: TAK-925 — TAK-925
  Arms: Cohort A'1; TAK-925 (Dose Level A'1); Cohort A'2; TAK-925 (Dose Level A'2); Cohort A1; TAK-925 (Dose Level A1); Cohort A2; TAK-925 (Dose Level A2); Cohort A3; TAK-925 (Dose Level A3); Cohort A4; TAK-925 (Dose Level A4); Cohort A5; TAK-925 (Dose Level A5); Cohort A6; TAK-925 (Dose Level A6); Cohort B1; TAK-925 (Dose Level B1); Cohort B2; TAK-925 (Dose Level B2); Cohort B3; TAK-925 (Dose Level B3); Cohort B4; TAK-925 (Dose Level B4); Cohort C1; TAK-925 (Dose Level C1); Cohort C2; TAK-925 (Dose Level C2)
Drug: Placebo — TAK-925 Placebo
  Arms: Part A (Cohorts A1-A6); TAK-925 Placebo; Part B (Cohorts B1-B4); TAK-925 Placebo; Part C (Cohorts C1-C2); TAK-925 Placebo

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of TAK-925 when administered to healthy participants and narcolepsy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-925. TAK-925 is being tested in healthy participants and participants with narcolepsy. This study will look at the safety, tolerability, pharmacokinetics, and efficacy of TAK-925.

This study will consist of three parts. Part A will be a randomized, double-blind, placebo-controlled, multiple rising dose (MRD) study in healthy participants. Part B is a randomized, double-blind, placebo-controlled MRD study in participants with narcolepsy. Part C is a randomized, double-blind, placebo-controlled, parallel group, multiple repeat dose study in participants with narcolepsy. Part A' is a single dose study in healthy participants.

The study will enroll approximately 96 participants planned as total. All participants except Part A' will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the participants and study doctor during the study (unless there is an urgent medical need):

Part A:

* TAK-925 (Dose Levels A1-A6)
* Placebo

Part B:

* TAK-925 (Dose Levels B1-B4)
* Placebo

Part C:

* TAK-925 (Dose Levels C1-C2)
* Placebo

Part A':

• TAK-925 (Dose Levels A'1-A'2)

All participants will be asked to take TAK-925 or Placebo at the same time each day from Day 1 to Day 7 in Parts A, B and C, and take TAK-925 on Day 1 in Part A'.

This multi-center trial will be conducted in Japan. The overall study period is approximately 15 days in Parts A, B and C, and approximately 7 days for Part A'. Participants will be partly admitted to a hospital during the study.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult participants and Healthy elderly participants:

• Participant weighs at least 50 kg (Healthy adults participants) / 40 kilogram (kg) (Healthy elderly participants) and has a body mass index (BMI) from 18.5 to 30 kilogram per square meter (kg/m^2), inclusive at Screening.

Narcolepsy participants:

* Participants weighs at least 40 kg inclusive at Screening (>=50 kg is required for Cohort B4).
* A diagnosis of narcolepsy, as defined by the International Classification of Sleep Disorders, Third Edition (ICSD-3).
* At Day -1, Epworth sleepiness scale (ESS) score >=10

Exclusion Criteria:

All Participants:

* Participants consume excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
* Participants have a moderate to severe substance use disorder.
* Participants have a risk of suicide according to endorsement of item 4 or 5 with Screening/Baseline visit C-SSRS (Columbia Suicide Severity Rating Scale) or has made a suicide attempt in the previous 6 months.
* Participants have a lifetime history of major psychiatric disorder, such as bipolar disorder or schizophrenia.
* Participants experienced sleep wake cycle disturbance with external factors such as irregular work hours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (3):
- Japan (3):
  - Sumida Hospital, Sumida-ku, Tokyo
  - Hakata Clinic, Fukuoka
  - PS Clinic, Fukuoka

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in Japan from 21 November 2018 to 24 October 2019.
Pre-assignment Details: Healthy participants were enrolled in Part A and A' (exploratory), NT1 in Part B and NT2 in Part C, to receive TAK-925 multiple rising dose of 44 mg (milligram), 112 mg,180 mg or placebo in Part A, 11 mg, 44 mg or placebo in Part B, multiple dose of TAK-925 44 mg, 112 mg or placebo in Part C.
Groups:
- Part A, Cohorts A1-A3: Pooled Placebo: TAK-925 placebo-matching, infusion, intravenously, once daily from Day 1 through Day 7 in healthy participants.
- Part A, Cohort A1: TAK-925 44 mg: TAK-925 44 mg, infusion, intravenously, once daily from Day 1 through Day 7 in healthy participants.
- Part A, Cohort A2: TAK-925 112 mg: TAK-925 112 mg, infusion, intravenously, once daily from Day 1 through Day 7 in healthy participants.
- Part A, Cohort A3: TAK-925 180 mg: TAK-925 180 mg, infusion, intravenously, once daily from Day 1 through Day 7 in healthy participants.
- Part B, Cohorts B1-B2: Pooled Placebo: TAK-925 placebo-matching, infusion, intravenously, once daily from Day 1 through Day 7 in narcolepsy type 1 (NT1) participants.
- Part B, Cohort B1: TAK-925 11 mg: TAK-925 11 mg, infusion, intravenously, once daily from Day 1 through Day 7 in NT1 participants.
- Part B, Cohort B2: TAK-925 44 mg: TAK-925 44 mg, infusion, intravenously, once daily from Day 1 through Day 7 in NT1 participants.
- Part C, Cohorts C1-C2: Pooled Placebo: TAK-925 placebo-matching, infusion, intravenously, once daily from Day 1 through Day 7 in narcolepsy type 2 (NT2) participants.
- Part C, Cohort C1: TAK-925 44 mg: TAK-925 44 mg, infusion, intravenously, once daily from Day 1 through Day 7 in NT2 participants.
- Part C, Cohort C2: TAK-925 112 mg: TAK-925 112 mg, infusion, intravenously, once daily from Day 1 through Day 7 in NT2 participants.
- Part A', Cohort A'1: TAK-925 112 mg: TAK-925 112 mg, solution, orally, once on Day 1 in healthy participants.
Period: Overall Study
Arm/Group | Part A, Cohorts A1-A3: Pooled Placebo | Part A, Cohort A1: TAK-925 44 mg | Part A, Cohort A2: TAK-925 112 mg | Part A, Cohort A3: TAK-925 180 mg | Part B, Cohorts B1-B2: Pooled Placebo | Part B, Cohort B1: TAK-925 11 mg | Part B, Cohort B2: TAK-925 44 mg | Part C, Cohorts C1-C2: Pooled Placebo | Part C, Cohort C1: TAK-925 44 mg | Part C, Cohort C2: TAK-925 112 mg | Part A', Cohort A'1: TAK-925 112 mg
Started | 6 | 6 | 6 | 6 | 4 | 4 | 5 | 5 | 4 | 5 | 6
Completed | 6 | 6 | 6 | 6 | 4 | 4 | 5 | 5 | 4 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set was defined as all participants who received at least one dose of study drug.
Groups:
- Part B, Cohorts B1-B2: Pooled Placebo: TAK-925 placebo-matching, infusion, intravenously, once daily from Day 1 through Day 7 in NT1 participants.
- Part C, Cohorts C1-C2: Pooled Placebo: TAK-925 placebo-matching, infusion, intravenously, once daily from Day 1 through Day 7 in NT2 participants.
- Total: Total of all reporting groups
Arm/Group | Part A, Cohorts A1-A3: Pooled Placebo | Part A, Cohort A1: TAK-925 44 mg | Part A, Cohort A2: TAK-925 112 mg | Part A, Cohort A3: TAK-925 180 mg | Part B, Cohorts B1-B2: Pooled Placebo | Part B, Cohort B1: TAK-925 11 mg | Part B, Cohort B2: TAK-925 44 mg | Part C, Cohorts C1-C2: Pooled Placebo | Part C, Cohort C1: TAK-925 44 mg | Part C, Cohort C2: TAK-925 112 mg | Part A', Cohort A'1: TAK-925 112 mg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 4 | 5 | 5 | 4 | 5 | 6 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.8 (4.71) | 24.7 (3.88) | 23.8 (3.54) | 22.3 (0.52) | 28.3 (9.18) | 38.0 (3.92) | 27.6 (8.20) | 31.8 (11.14) | 31.3 (7.50) | 25.0 (5.87) | 21.7 (2.88) | 26.6 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 3 | 3 | 2 | 0 | 13
  Male | 6 | 6 | 6 | 6 | 3 | 2 | 3 | 2 | 1 | 3 | 6 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 6 | 6 | 6 | 6 | 4 | 4 | 5 | 5 | 4 | 5 | 6 | 57
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m˄2)] | 22.42 (0.968) | 21.12 (1.030) | 22.37 (1.960) | 21.87 (2.360) | 24.83 (2.378) | 27.33 (4.955) | 24.68 (4.791) | 20.88 (3.565) | 22.83 (4.213) | 22.18 (3.489) | 21.05 (1.174) | 22.66 (3.210)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 170.2 (4.71) | 173.3 (4.84) | 168.8 (5.85) | 170.8 (4.71) | 169.8 (7.80) | 165.3 (8.18) | 166.8 (7.56) | 162.2 (5.02) | 158.0 (5.60) | 164.6 (5.46) | 170.7 (3.44) | 167.8 (6.63)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 64.58 (5.486) | 62.75 (3.250) | 63.72 (7.392) | 63.60 (7.987) | 72.90 (13.071) | 75.20 (18.150) | 70.32 (15.554) | 56.20 (11.689) | 57.73 (13.072) | 61.68 (10.055) | 60.60 (4.549) | 64.14 (10.706)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE was defined as an AE with an onset that occurs after receiving study drug.
Time Frame: From the first dose of study drug up to 7 days after the last dose of study drug (up to Day 15)
Population: The safety set was defined as all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Cohorts A1-A3: Pooled Placebo | Part A, Cohort A1: TAK-925 44 mg | Part A, Cohort A2: TAK-925 112 mg | Part A, Cohort A3: TAK-925 180 mg | Part B, Cohorts B1-B2: Pooled Placebo | Part B, Cohort B1: TAK-925 11 mg | Part B, Cohort B2: TAK-925 44 mg | Part C, Cohorts C1-C2: Pooled Placebo | Part C, Cohort C1: TAK-925 44 mg | Part C, Cohort C2: TAK-925 112 mg | Part A', Cohort A'1: TAK-925 112 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 4 | 5 | 5 | 4 | 5 | 6
Participants | 1 | 0 | 2 | 4 | 1 | 1 | 5 | 0 | 1 | 3 | 0

2. Secondary Outcome: Parts A, B and C; Ceoi: Observed Plasma Concentration at the End of Infusion for TAK-925
Description: This assessment was pre-specified to be conducted for participants in "Part A', Cohort A'1: TAK-925 112 mg" as exploratory measures.
Time Frame: Part A,Days 1,7:pre-infusion(inf),0.5,1, 1.5, 2, 4, 6, 8, 9 hours(h)post start of inf;0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 6, 10, 15 h post end of inf;Part B,C:Days 1,7:Pre-inf, 1, 2, 4, 6, 9 h post start of inf; 0.17, 0.5, 2, 6, 10, 15 h post end of inf
Population: The pharmacokinetic (PK) set was defined as all participants who received at least one dose of study drug and provided sufficient PK measurements available to estimate PK parameters, at least 1 estimable PK parameter.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A, Cohort A1: TAK-925 44 mg | Part A, Cohort A2: TAK-925 112 mg | Part A, Cohort A3: TAK-925 180 mg | Part B, Cohort B1: TAK-925 11 mg | Part B, Cohort B2: TAK-925 44 mg | Part C, Cohort C1: TAK-925 44 mg | Part C, Cohort C2: TAK-925 112 mg
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 5 | 4 | 5
nanogram per milliliter (ng/mL)
  Day 1 | 74.49 (4.3433) | 166.9 (20.995) | 300.2 (50.532) | 17.39 (1.2842) | 70.20 (18.798) | 68.74 (7.3623) | 156.1 (29.210)
  Day 7 | 70.31 (8.4434) | 159.2 (23.560) | 295.5 (46.173) | 17.68 (1.7176) | 73.20 (14.980) | 70.87 (7.4375) | 153.9 (24.876)

3. Secondary Outcome: Parts A, B and C; AUCtau: Area Under the Plasma Concentration-Time Curve During a Dosing Interval for TAK-925
Description: as for outcome 2
Time Frame: as for outcome 2
Population: The PK set was defined as all participants who received at least one dose of study drug and provided sufficient PK measurements available to estimate PK parameters, at least 1 estimable PK parameter.
Measure: Geometric Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part A, Cohort A1: TAK-925 44 mg | Part A, Cohort A2: TAK-925 112 mg | Part A, Cohort A3: TAK-925 180 mg | Part B, Cohort B1: TAK-925 11 mg | Part B, Cohort B2: TAK-925 44 mg | Part C, Cohort C1: TAK-925 44 mg | Part C, Cohort C2: TAK-925 112 mg
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 5 | 4 | 5
hour*nanogram per milliliter (h*ng/mL)
  Day 1 | 662.4 (70.718) | 1516 (151.45) | 2615 (392.89) | 164.2 (18.257) | 682.3 (126.81) | 648.3 (80.748) | 1496 (279.16)
  Day 7 | 650.7 (78.156) | 1523 (174.40) | 2747 (372.96) | 182.7 (22.603) | 722.7 (102.28) | 657.1 (72.833) | 1519 (248.46)

4. Secondary Outcome: Parts A, B and C; Rac (AUC): Accumulation Ratio Based on AUCtau for TAK-925
Description: Accumulation Ratio of AUC was calculated as AUCtau on Day 7 divided by AUCtau on Day 1. This assessment was pre-specified to be conducted for participants in "Part A', Cohort A'1: TAK-925 112 mg" as exploratory measures.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part A, Cohort A1: TAK-925 44 mg | Part A, Cohort A2: TAK-925 112 mg | Part A, Cohort A3: TAK-925 180 mg | Part B, Cohort B1: TAK-925 11 mg | Part B, Cohort B2: TAK-925 44 mg | Part C, Cohort C1: TAK-925 44 mg | Part C, Cohort C2: TAK-925 112 mg
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 5 | 4 | 5
ratio | 0.9832 (0.041034) | 1.009 (0.080171) | 1.050 (0.020000) | 1.118 (0.14637) | 1.062 (0.066062) | 1.017 (0.098127) | 1.018 (0.030760)

5. Secondary Outcome: Parts B and C: Change From Baseline in Sleep Latency in the Maintenance of Wakefulness Test (MWT) at Days 1 and 7
Description: The MWT is a validated objective measure that is used to measure excessive daytime sleepiness in clinical studies. It has been used as a secondary outcome measure for excessive daytime sleepiness. The MWT evaluates a person's ability to remain awake under soporific conditions for a defined period of time. Wakefulness in this study was measured indirectly by time to fall asleep using MWT. In this study, four 40-minute (1 session) MWT assessments per day was administered on Baseline, Day 1 and Day 7. MWT sleep latency ranges from 0 to 40 minutes, with longer sleep latency indicating greater ability to stay awake.
Time Frame: Baseline, Day 1 and Day 7
Population: The pharmacodynamic (PD) set was defined as all participants who received at least one dose of study drug. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part B, Cohorts B1-B2: Pooled Placebo | Part B, Cohort B1: TAK-925 11 mg | Part B, Cohort B2: TAK-925 44 mg | Part C, Cohorts C1-C2: Pooled Placebo | Part C, Cohort C1: TAK-925 44 mg | Part C, Cohort C2: TAK-925 112 mg
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 4 | 5
minutes
  Baseline: number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 5
  Baseline | 1.97 (0.850) | 2.03 (0.717) | 5.23 (4.029) | 4.13 (3.280) | 6.83 (3.924) | 7.33 (5.932)
  Change at Day 1: number analyzed (Participants) | 4 | 4 | 4 | 5 | 3 | 5
  Change at Day 1 | -0.66 (0.892) | 35.13 (4.268) | 34.19 (4.398) | 2.58 (3.751) | 23.88 (2.955) | 31.15 (5.507)
  Change at Day 7: number analyzed (Participants) | 4 | 4 | 5 | 5 | 3 | 5
  Change at Day 7 | -0.38 (0.621) | 21.00 (12.141) | 34.78 (4.029) | 2.35 (3.369) | 25.79 (7.544) | 28.28 (4.886)
Statistical Analysis 1: Comparison: Part B, Cohorts B1-B2: Pooled Placebo vs Part B, Cohort B1: TAK-925 11 mg; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — P-value was obtained using MMRM analysis. The p-value for each treatment group is for the comparison of that treatment group to the placebo treatment group on Day 1
Statistical Analysis 2: Comparison: Part B, Cohorts B1-B2: Pooled Placebo vs Part B, Cohort B2: TAK-925 44 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Part B, Cohorts B1-B2: Pooled Placebo vs Part B, Cohort B1: TAK-925 11 mg; Test type: Superiority; p = 0.0002, MMRM — P-value was obtained using MMRM analysis. The p-value for each treatment group is for the comparison of that treatment group to the placebo treatment group on Day 7
Statistical Analysis 4: Comparison: Part B, Cohorts B1-B2: Pooled Placebo vs Part B, Cohort B2: TAK-925 44 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 3]
Statistical Analysis 5: Comparison: Part C, Cohorts C1-C2: Pooled Placebo vs Part C, Cohort C1: TAK-925 44 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Part C, Cohorts C1-C2: Pooled Placebo vs Part C, Cohort C2: TAK-925 112 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Part C, Cohorts C1-C2: Pooled Placebo vs Part C, Cohort C1: TAK-925 44 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 3]
Statistical Analysis 8: Comparison: Part C, Cohorts C1-C2: Pooled Placebo vs Part C, Cohort C2: TAK-925 112 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 3]

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events (AEs) that started after the first dose of study drug up to 7 days after the last dose of study drug (up to Day 15)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part A, Cohorts A1-A3: Pooled Placebo | Part A, Cohort A1: TAK-925 44 mg | Part A, Cohort A2: TAK-925 112 mg | Part A, Cohort A3: TAK-925 180 mg | Part B, Cohorts B1-B2: Pooled Placebo | Part B, Cohort B1: TAK-925 11 mg | Part B, Cohort B2: TAK-925 44 mg | Part C, Cohorts C1-C2: Pooled Placebo | Part C, Cohort C1: TAK-925 44 mg | Part C, Cohort C2: TAK-925 112 mg | Part A', Cohort A'1: TAK-925 112 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/4 | 0/5 | 0/5 | 0/4 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/4 | 0/5 | 0/5 | 0/4 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 2/6 | 4/6 | 1/4 | 1/4 | 5/5 | 0/5 | 1/4 | 3/5 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Cohorts A1-A3: Pooled Placebo (N=6) | Part A, Cohort A1: TAK-925 44 mg (N=6) | Part A, Cohort A2: TAK-925 112 mg (N=6) | Part A, Cohort A3: TAK-925 180 mg (N=6) | Part B, Cohorts B1-B2: Pooled Placebo (N=4) | Part B, Cohort B1: TAK-925 11 mg (N=4) | Part B, Cohort B2: TAK-925 44 mg (N=5) | Part C, Cohorts C1-C2: Pooled Placebo (N=5) | Part C, Cohort C1: TAK-925 44 mg (N=4) | Part C, Cohort C2: TAK-925 112 mg (N=5) | Part A', Cohort A'1: TAK-925 112 mg (N=6)
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03748979/SAP_000.pdf
  • Study Protocol (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT03748979/Prot_001.pdf